CLINICAL TRIAL: NCT01494311
Title: Lidocaine/Tetracaine Patch (Rapydan) for Topical Anaesthesia Before Arterial Access: A Double-blind, Randomized Trial
Brief Title: Rapydan Topical Anaesthesia for Arterial Cannulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: The Cleveland Clinic (Other); Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Kurt Rutzler, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2010/1046
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Arterial Catheterization
Keywords: Arterial catheter; arterial cannula; Rapydan; lidocaine/tetracaine patch; topical anaesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo patch and lidocaine injection (Active Comparator): Fourty-five patients were randomly assigned to receive a placebo patch, looking identically to the Rapydan patch and subsequent subcutaneous injection of 0.5 ml of lidocaine 1%.
  Interventions: Drug: Placebo Patch; Drug: Subcutaneous injection of 0.5 ml Lidocain 1%
- Lidocaine/tetracaine patch (Experimental): Fourty-five patients were randomly assigned to receive a lidocaine/tetracaine patch, followed by subcutaneous injection 0.5 ml of normal saline solution.
  Interventions: Drug: Lidocaine/tetracaine patch; Drug: Subcutaneous injection of saline

INTERVENTIONS:
Drug: Lidocaine/tetracaine patch — The lidocaine/tetracaine patch topical anesthetic patch contains 70 mg each of lidocaine and tetracaine. The central area of each patch consists of a Controlled Heat Assisted Drug Delivery pod which is designed to warm the skin to 26-34°C, theoretically enhancing drug absorption and allowing application just 20 minutes before percutaneous procedures. A active or placebo patch was placed on each patient's wrist in the region of the maximum radial artery pulsation. After 20 minutes, the patch was removed.
  Other Names: Rapydan; Synera, 76667213
  Arms: Lidocaine/tetracaine patch
Drug: Placebo Patch — A placebo patch was placed on each patient's wrist in the region of the maximum radial artery pulsation. After 20 minutes, the patch was removed.
  Arms: Placebo patch and lidocaine injection
Drug: Subcutaneous injection of 0.5 ml Lidocain 1% — After removing the patch, a blinded investigator injected 0.5 ml of 1% lidocaine solution. Three minutes after injection, an attempt was made to cannulate the radial artery with a 20-gauge catheter.
  Arms: Placebo patch and lidocaine injection
Drug: Subcutaneous injection of saline — After removing the patch, a blinded investigator injected 0.5 ml saline solution. Three minutes after injection, an attempt was made to cannulate the radial artery with a 20-gauge catheter.
  Arms: Lidocaine/tetracaine patch

SUMMARY:
Arterial catheterization is painful and is associated with patient stress and anxiety. Analgesia is usually provided by subcutaneous injection of local anesthetic. An alternative is topical anaesthesia, such as Rapydan which is a novel topical anesthetic patch containing 70 mg each of lidocaine and tetracaine. We therefore tested the hypothesis that Rapydan patch analgesia is non-inferior to subcutaneous local anesthetic.

DETAILED DESCRIPTION:
Many clinical procedures including arterial and venous punctures, percutaneous venous catheter insertion, lumbar puncture, and dermatological procedures are associated with pain and consequent patient discomfort.1-2 With the exception of venopuncture, arterial puncture is the most common invasive procedure performed on critically ill patients. Also, it is often necessary before induction of anaesthesia for invasive measurements of blood pressure and collection of arterial blood samples in patients undergoing major cardiac surgery. Injection of local anesthetics before insertion causes intra-dermal turgor and can trigger local vasoconstriction, both of which reduce puncture success rate.

An alternative approach is to use topical anesthesia for percutaneous procedures. However, intact skin presents a significant barrier to topical anesthetic preparations. Therefore, topical anesthetic preparations typically must be applied under occlusive dressings for 45-60 minutes before vascular access - which is often longer than is clinically practical.

Rapydan (also known as Synera in the United States) is a novel topical anesthetic patch that contains 70 mg each of lidocaine and tetracaine. The central area of each Rapydan patch consists of a Controlled Heat Assisted Drug Delivery pod which is designed to allow for application just 20 minutes before percutaneous procedures. However, the efficacy of Rapydan topical analgesia has yet to be quantified for the more intense pain resulting from arterial puncture. We thus compared routine analgesia (subcutaneous injection with 0.5 ml of 1% lidocaine) with heated lidocaine/tetracaine patches. Specifically, we tested the hypothesis that lidocaine/tetracaine patch analgesia is non-inferior to that provided by subcutaneous lidocaine injection for insertion of arterial catheters.

Ninty patients undergoing elective major cardiac surgery were included in this prospective, double blind clinical trial. Patients were randomly assigned to receive either a lidocaine/tetracaine patch, followed by subcutaneous injection 0.5 ml of normal saline solution or placebo patch, looking identically to the Rapydan patch and subsequent subcutaneous injection of 0.5 ml of lidocaine 1%. Pain during arterial catheterization using 100-mm-long visual analog scale (VAS) was the primary outcome. Other outcomes were pain during anesthetic/saline injection and plasma tetracaine concentrations.

VAS pain scores during arterial puncture were comparable in both groups and Rapydan was non-inferior to subcutaneous lidocaine. Pain scores at the time of subcutaneous injection were significantly lower (better) in patients assigned to the lidocaine/tetracaine patch than to lidocaine (P = 0.001). Plasma tetracaine concentrations never exceeded the detection limit of 25 ng/ml at any time in any patient.

Both the lidocaine/tetracaine patch and subcutaneous injection of lidocaine provided comparable pain control during arterial catheter insertion. Subcutaneous lidocaine caused discomfort during injection whereas the lidocaine/tetracaine patch required placement 20 minutes before the procedure. Given adequate time, the patch provided better overall analgesia by obviating the need for subcutaneous infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Patients having elective valve-replacement or coronary artery bypass grafting requiring arterial access before induction of anaesthesia.

Exclusion Criteria:

* analgesic use within 24 hours before surgery
* injury or infection at the planned puncture site
* known allergy to local anesthetics
* drug abuse
* alcoholism or psychiatric disorders
* childbearing potential without adequate birth control
* abnormal Allen's test

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pain during arterial catheterization | During and minutes after arterial cannula insertion, day 1.
  After finishing the puncture procedure, patients were asked to rate their worst pain during subcutaneous injection, during insertion of arterial cannula, and one minute after catheter insertion using a 100-mm-long visual analog scale (VAS). The use of a VAS to measure pain and discomfort has been validated in the several settings of chronic pain, acute postoperative pain, and acute non-surgical pain.

SECONDARY OUTCOMES:
Pain during annethetic/saline injection. | During and minutes after injection, day 1.
  After finishing the puncture procedure, patients were asked to rate their worst pain during subcutaneous injection, during insertion of arterial cannula, and one minute after catheter insertion using a 100-mm-long visual analog scale (VAS).
Blood concentration of plasma tetracaine | Minutes before and after patch application, day 1.
  Blood for measurement of plasma tetracaine concentrations sampled: 1) before patch application; 2) 15 minutes after patch application; 3) immediately after successful arterial puncture; 4) 30 minutes after patch application; and, 5) 60 minutes after patch application. Only blood samples from patients assigned to the tetracaine/lidocaine patch were analyzed.
Patient Satisfaction | At conclusion of procedure, day 1.
  Patients also subjectively rated their procedure-related satisfaction on a four-point scale: 0 = unsatisfied; 1 = moderately satisfied; 2 = satisfied; and, 3 = very satisfied.
Investigator's evaluatuion of pain during catheter insertion | At conclusion of procedure, day 1.
  Investigators who were unaware of the randomization estimated each patient's pain intensity at the time of catheter insertion on a four-point scale with 0 indicating no pain and 3 indicating severe pain.
Difficulty of puncture | During catheter insertion, day 1.
  The difficulty of the puncture was assessed using a 5-point scale with 1 being insertion at first attempt through 5 which indicated failure to insert the catheter.
Number of punctrue attempts | During catheter insertion, day 1.
  The number of puncture attempts were documented by the investigator.
Incidence of edema and erthema at the patch site | Evaluated immediately after patch removed, day 1.
  After the patches were removed an investigator, blinded to the study randomization, evaluated the treatment sites for skin reactions including edema and erythema using a 5-point Likert scale (1 = none; 5 = vigorous).

CONTACTS AND LOCATIONS:
Locations (3):
- Cleveland Clinic Department of Outcomes Research, Cleveland, Ohio, United States
- Medical University of Vienna, Vienna, Austria
- Population Health Research Institute, McMaster University, Hamilton, Ontario, Canada